CLINICAL TRIAL: NCT06337058
Title: The Effect of Motivational Interviews With Women Experiencing Sexual Dysfunction During Menopause on Quality of Sexual Life and Self-Efficacy
Brief Title: Motivational Interviews With Women Experiencing Sexual Dysfunction During Menopause Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hülya KAMALAK (Other)
Responsible Party: Sponsor-Investigator, Hülya KAMALAK, Lecturer, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KSUHULYAKAMALAK001
Record Dates: First submitted 2024-03-01; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Sexual Dysfunction
Keywords: Menopause Period; Motivational Interview; Sexual Dysfunction; Sexual Quality of Life; Midwifery
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): intervention group
  Interventions: Behavioral: Experimental group (motivational interview)
- control group (No Intervention): control group

INTERVENTIONS:
Behavioral: Experimental group (motivational interview) — For the menopausal women with sexual dysfunction in the experimental group, pre-test data were obtained by applying the 'Personal Information Form', the 'Sexual Quality of Life Scale-Woman' and the 'Sexual Self-Efficacy Scale' before starting the motivational interviews. After the pre-test data were obtained, a total of 4 sessions of motivational interviews were provided, one session per week for four weeks. At the end of four weeks, post-test data were obtained by applying the "Arizona Sexual Experiences Scale", "Sexual Quality of Life Scale-Women" and "Sexual Self-Efficacy Scale".
  The researcher received a training on motivational interview techniques before implementing the intervention for menopausal women in the experimental group.
  Arms: experimental group

SUMMARY:
The aim of this study is to evaluate the effect of motivational interviews with women who experience sexual dysfunction during menopause on sexual quality of life and self-efficacy.The population of the study consisted of menopausal women who applied to the gynecology outpatient clinic of Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital. It was calculated as 164 women (82 experimental, 82 control).In data collection, 'Personal Information Form (EK- )', 'Arizona Sexual Experiences Scale (ACYÖ) (EK- )', 'Sexual Quality of Life Scale-Female (SIQQ-F) (EK-)' and 'Sexual Self-Efficacy Scale' (Annex- )' was used.

DETAILED DESCRIPTION:
Aim: This study was conducted to determine the effect of motivational interviewing on sexual quality of life and sexual self-efficacy in menopausal women with sexual dysfunction.

Methods: This randomized controlled study was conducted with 164 menopausal women with sexual dysfunction who applied to the gynecology outpatient clinic of a university hospital in southern Turkey (82 experimental, 82 control). The data were collected using a personal information form, the Arizona Sexual Experiences Scale - Female Version Questionnaire (ASEX-F), the Sexual Quality of Life-Female Questionnaire (SQOL-F) and the Sexual Self-Efficacy Scale (SSES). Menopausal women with sexual dysfunction (with a score of 19 and above on the ASEX-F) who applied to the gynecology outpatient clinic of the relevant hospital were invited to the study.

Before starting the motivational interviews with menopausal women in the experimental group; the PIF, the SQOL-F and the SSES were applied and their pre-test data were obtained. After the pre-test data were obtained, 4 sessions of motivational interviews were conducted with the women, 1 session per week for four weeks. Motivational interviews were completed with face-to-face interviews lasting 20-30 minutes for each woman, and those in the control group did not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being able to read and write,
* Ability to communicate
* Being sexually active,
* Having entered menopause in the last 3 years,
* Having entered menopause naturally,
* Diagnosis of sexual dysfunction according to the Arizona Sexual Experiences Scale (total score ≥19).

Exclusion Criteria:

* Having any diagnosed psychiatric illness,
* Having entered menopause surgically,
* Being on hormone replacement therapy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Arizona Sexual Experiences Scale - Female Version Questionnaire (ASEX-F) | 1 day At the first interview, the Arizona Sexual Experiences Scale - Female Version Survey (ASEX-F) was administered to menopausal women in both groups as a pretest.
  This Likert-type self-assessment scale, available in both female and male forms, consists of five items. Its internal consistency and reliability (Cronbach's alpha) values ranged from 0.89 to 0.90. It has been determined to be useful for detecting sexual dysfunction. Each item on the scale is scored from 1 to 6, with a total score ranging from 5 to 30. A total score of 19 or higher, any item scoring 5 or 6 points, or four or more items scoring 4 points indicate the presence of sexual dysfunction. Low scores represent an effective, comfortable, and satisfactory sexual response, while high scores indicate the presence of sexual dysfunction.
Arizona Sexual Experiences Scale - Female Version Questionnaire (ASEX-F) | Four week after the first interview, the Arizona Sexual Experiences Scale - Female Version Survey (ASEX-F) was applied to all menopausal women in all two groups as a posttest
  This Likert-type self-assessment scale, available in both female and male forms, consists of five items. Its internal consistency and reliability (Cronbach's alpha) values ranged from 0.89 to 0.90. It has been determined to be useful for detecting sexual dysfunction. Each item on the scale is scored from 1 to 6, with a total score ranging from 5 to 30. A total score of 19 or higher, any item scoring 5 or 6 points, or four or more items scoring 4 points indicate the presence of sexual dysfunction. Low scores represent an effective, comfortable, and satisfactory sexual response, while high scores indicate the presence of sexual dysfunction.
Sexual Quality of Life-Female Questionnaire (SQOL-F) | 1 day At the first interview, the Sexual Quality of Life-Female Questionnaire (SQOL-F) was administered to menopausal women in both groups as a pretest.
  The scale consists of a total of 18 items, requiring responses regarding sexual problems in the last 4 weeks. This is a Likert-type scale with six response options. For item scoring from 0 to 5, the minimum and maximum possible scores on the scale are 0 and 90, respectively. For item scoring between 1 and 6, the minimum and maximum possible scores on the scale are 18 and 108, respectively. In this study, the scoring system between 1 and 6 was used. Higher scores on the scale indicate a good quality of sexual life.
Sexual Quality of Life-Female Questionnaire (SQOL-F) | Four week after the first interview, the Sexual Quality of Life-Female Questionnaire (SQOL-F) was applied to all menopausal women in all two groups as a posttest
  The scale consists of a total of 18 items, requiring responses regarding sexual problems in the last 4 weeks. This is a Likert-type scale with six response options. For item scoring from 0 to 5, the minimum and maximum possible scores on the scale are 0 and 90, respectively. For item scoring between 1 and 6, the minimum and maximum possible scores on the scale are 18 and 108, respectively. In this study, the scoring system between 1 and 6 was used. Higher scores on the scale indicate a good quality of sexual life.
Sexual Self-Efficacy Scale (SSES) | 1 day At the first interview, the Sexual Self-Efficacy Scale (SSES) was administered to menopausal women in both groups as a pretest.
  The SSES was developed by Humphreys and Kennett (2010), and its Turkish validity and reliability study was conducted by Çelik (2012). The 8-point Likert scale consists of 5 items, scoring from 1 = Strongly Disagree to 8 = Strongly Agree and representing a single factor. The self-reporting scale was developed to determine individuals' sexual self-efficacy, where total scores are obtained by reverse coding items 3 and 4. Higher scores on the scale indicate higher levels of sexual self-efficacy. Total scale score ranges between 5 and 40.The Cronbach's alpha coefficient for the scale is 0.71. In this study, the Cronbach's alpha reliability coefficient was found as 0.93 for the experimental group and 0.90 for the control group.
Sexual Self-Efficacy Scale (SSES) | Four week after the first interview, the Sexual Self-Efficacy Scale (SSES) was applied to all menopausal women in all two groups as a posttest
  The SSES was developed by Humphreys and Kennett (2010), and its Turkish validity and reliability study was conducted by Çelik (2012). The 8-point Likert scale consists of 5 items, scoring from 1 = Strongly Disagree to 8 = Strongly Agree and representing a single factor. The self-reporting scale was developed to determine individuals' sexual self-efficacy, where total scores are obtained by reverse coding items 3 and 4. Higher scores on the scale indicate higher levels of sexual self-efficacy. Total scale score ranges between 5 and 40.The Cronbach's alpha coefficient for the scale is 0.71. In this study, the Cronbach's alpha reliability coefficient was found as 0.93 for the experimental group and 0.90 for the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya KAMALAK, Phd, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutçu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No